CLINICAL TRIAL: NCT01448902
Title: A Study Of The Effects Of OC000459 On Responses To Allergen Challenge In The Vienna Chamber In Subjects Known To Suffer From Grass Pollen Induced Allergic Rhinitis
Brief Title: A Study Of The Effects Of OC000459 In Subjects Known To Suffer From Grass Pollen Induced Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oxagen Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: OC000459/007/06; 2007-000017-11 (EudraCT Number)
Record Dates: First submitted 2011-07-27; First posted 2011-10-07 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-10

CONDITIONS: Allergic Rhinitis
Keywords: Allergic rhinitis; CRTH2
MeSH Terms: conditions — Rhinitis, Allergic | interventions — (5-fluoro-2-methyl-3-quinolin-2-ylmethylindo-1-yl)acetic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- OC000459 (Experimental)
  Interventions: Drug: OC000459
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OC000459 — OC000459 200mg bid for 8 days
  Arms: OC000459
Drug: Placebo — Placebo bid for 8 days
  Arms: Placebo

SUMMARY:
The study will assess the efficacy of OC000459 200 mg twice daily orally in comparison to placebo when subjects are challenged in the Vienna Challenge Chamber for 6 hours. This is a randomised, double blind, placebo controlled, two way crossover evaluation. There will be a screening period of up to three weeks and a washout period of at least one week between the two treatment periods. There will be a follow up one to three weeks after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18 to 50 years with a history of symptoms of grass pollen related allergic rhinitis within the previous two years.
* Subjects must be free from significant cardiac, pulmonary, gastrointestinal, hepatic, renal, haematological, neurological and psychiatric disease as determined by history, physical examination and screening investigations.
* FEV1 within normal limits (≥90% of predicted).
* Atopy defined by a positive cutaneous response to mixed grass pollen within the last 12 months or at screening.
* Asymptomatic at screening
* Non smokers for at least the past 12 months

Exclusion Criteria:

* Medical conditions likely to affect the outcome of the study.
* Nasal conditions likely to affect the outcome of the study, i.e. nasal septal perforations, nasal polyps, sinus disease, chronic nasal obstruction, or other nasal diseases.
* Presence of any respiratory disease other than a history of mild stable asthma not requiring treatment and associated with normal lung function
* Immunotherapy treatment course including inhaled or local corticosteroids in the past 28 days.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-03; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Efficacy of OC00045 on response to allergen challenge as measured by change in Total Nasal Symptom Score | 8 days
  To assess the efficacy of OC000459 200 mg twice daily orally in comparison to placebo when subjects are challenged in the Vienna Challenge Chamber for 6 hours as shown by the effect on Total Nasal Symptom Score

SECONDARY OUTCOMES:
OC000459 safety as determined by adverse events, laboratory parameters, lung function and vital signs | 8 days
  To assess the safety of this treatment schedule in male subjects with allergic rhinitis as assessed via adverse events, clinical chemistry and haematology, FEV1 and vital signs.
OC000459 plasma concentration (Cmin) | 8 days
  To assess plasma levels of OC000459 at the time of allergen challenge (trough plasma level).

CONTACTS AND LOCATIONS:
Overall Officials: Friedrich Horak, Prof Dr, Principal Investigator — Vienna Challenge Chamber
Locations (1):
- Vienna Challenge Chamber, Vienna, Austria

REFERENCES:
- [Derived] Horak F, Zieglmayer P, Zieglmayer R, Lemell P, Collins LP, Hunter MG, Steiner J, Lewis T, Payton MA, Perkins CM, Pettipher R. The CRTH2 antagonist OC000459 reduces nasal and ocular symptoms in allergic subjects exposed to grass pollen, a randomised, placebo-controlled, double-blind trial. Allergy. 2012 Dec;67(12):1572-9. doi: 10.1111/all.12042. Epub 2012 Oct 1. PMID 23025511